CLINICAL TRIAL: NCT04646590
Title: A Phase III Randomized, Double-blind, Placebo-controlled Clinical Trial in 18 Years of Age and Above to Determine the Safety and Efficacy of ZF2001, a Recombinant Novel Coronavirus Vaccine (CHO Cell) for Prevention of COVID-19
Brief Title: A Phase III Clinical Trial to Determine the Safety and Efficacy of ZF2001 for Prevention of COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2020-NCV-GJ01
Record Dates: First submitted 2020-11-25; First posted 2020-11-30 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Prevention of COVID-19; Safety and Efficacy
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Vaccine (Experimental): Recombinant Novel Coronavirus Vaccine (CHO cell), 0.5mL/vial, contains 25 μg NCP-RBD protein. After mixing, take all the liquid and inject intramuscularly into deltoid muscle of upper arm.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Placebo comparator (Placebo Comparator): Placebo for Recombinant Novel Coronavirus Vaccine (CHO cell), 0.5mL/vial, contains 0.25mg Aluminum hydroxide adjuvant. After mixing, take all the liquid and inject intramuscularly into deltoid muscle of upper arm.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) group — Intramuscular injection of deltoid muscle of upper armof 25μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Investigational Vaccine
Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group — Intramuscular injection of deltoid muscle of upper arm of 0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells) placebo.
  Arms: Placebo comparator

SUMMARY:
A randomized, double-blind, placebo-controlled international multicenter clinical trial design will be adopted. A total of 29,000 subjects aged 18 years and above are planned to be recruited, including 750 subjects aged 18-59 years and 250 subjects aged 60 years and above in China; 21,000 subjects aged 18-59 years and 7,000 subjects aged 60 years and above will be recruited outside China. Safety and immunogenicity will be evaluated among the Chinese subjects, and efficacy, immunogenicity and safety will be evaluated among the subjects outside China. Among them, 750 subjects aged 18-59 and 250 subjects aged 60 and above from outside China and all subjects from China will be selected as the immunogenicity subgroup for immunogenicity bridging study. The IgG levels of SARS-COV-2 neutralizing antibody and RBD protein binding antibody will be detected by blood sampling before vaccination, 14 days and 6 months after full course of vaccination to evaluate the immunogenicity and immune persistence.

DETAILED DESCRIPTION:
After signing the informed consent form, the volunteers aged 18 years and above will receive the relevant examinations after an inquiry by investigator of the medical history (including COVID-19 history), recent medication(vaccine) history, allergy history and concomitant medications, and demographic data collection by the investigators, including physical examination (skin and mucous membranes, lymph nodes, head, neck, chest, abdomen, spine/limbs), novel Coronavirus (SARS-COV-2) nucleic acid test and antibody test, urine pregnancy (women of childbearing age) test, and vital signs (blood pressure, axillary/oral temperature, pulse) evaluation.

Screening eligible subjects will be 1:1 randomly assigned to the experimental group and the placebo control group, and vaccinated as per the 0, 1, 2 month immunization schedule.

All adverse events (AEs) up to 30 minutes after each dose of vaccination, all AEs from 0 to 7 days (including both solicited and unsolicited), and all AES from 8 to 30 days (unsolicited) will be collected; All serious adverse events (SAEs) will be collected from the first dose of vaccination to 12 months after the whole vaccination.

The incidence rate and efficacy of any severity of COVID-9 of any severity 14 days after whole vaccination.

Blood samples (5ml) will be collected before the first dose of vaccination and 14 days and 6 months after the whole course of vaccination to detect neutralizing antibody of SARS-COV-2 and protein binding antibody IgG of receptor binding region (RBD) .

ELIGIBILITY:
Inclusion Criteria:

* Population aged 18 years and above;
* Subjects voluntarily participate in the study and sign the informed consent form; and are able to provide valid identification, and understand and comply with the requirements of the trial protocol;
* Female subjects of childbearing age agree to use effective contraceptive measures from the beginning of the study to 2 months after full course of vaccination.

Exclusion Criteria:

* Suspected or confirmed as fever(axillary temperature ≥37.3°C / oral temperature ≥37.5°C) within 72 hours before the enrollment, or axillary temperature ≥37.3°C / oral temperature ≥37.5°C at the day of screening;
* Diastolic blood pressure ≥ 100mmhg and / or systolic blood pressure ≥ 150mmhg;
* Patients with previous history of a COVID-19;
* Detection of SARS-COV-2 nucleic acid or antibody is positive;
* Those who are suffering from the following diseases:

  1. With thrombocytopenia, any coagulation dysfunction or receiving anti-coagulatory treatment
  2. Congenital or acquired immune deficiency or autoimmune disease history; no spleen, or history of splenic surgery and trauma, or receiving immunomodulator treatment within 6 months, e.g., immunosuppressive dose of glucocorticoids (reference dose: equivalent to 20mg/ day of prednisone, over 1 week); Or monoclonal antibodies; Or thymosin; Or interferon etc.; However, topical application (such as ointment, eye drops, inhalers or nasal sprays) is permitted;
  3. Symptoms related to acute respiratory tract infection (such as sneezing, nasal congestion, runny nose, cough, sore throat, loss of taste, chills, shortness of breath, etc.);
  4. Cancer patients (except basal cell carcinoma).
* With a history of serious allergy to any vaccine or any composition of Investigational product (including: aluminum preparations), such as allergic shock, allergic throat edema, allergic purpura, thrombocytopenic purpura, localized allergic necrosis reaction (Arthus reaction), dyspnea and angioneuroedema;
* Inoculated with subunit vaccine and inactivated vaccine within 14 days before the first dosing of investigational vaccine, or inoculated with attenuated live vaccine within 30 days;
* Previous receiving blood transfusion or blood relevant products (including immunoglobulin) within 3 months, or planning to receive such products from the starting of study to <6 months after the whole-course inoculation;
* Have participated in or are participating in other covid-19 related clinical trials;
* Women in breastfeeding period or in pregnant period (including women at childbearing age with positive result of urine pregnancy test);
* Considered by investigators as any disease or state possibly making the subject at unacceptable risk; not conforming to the requirements of study protocol; interference of assessment of reactions of vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28904 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The endpoint of efficacy study | 14 days to one year after whole vaccination
  The number of any severity of COVID-9 cases 14 days after whole vaccination
The endpoint of safety study | From the first dose of vaccination until 30 days after full course of vaccination
  Analysis of adverse events from the first dose of vaccination until 30 days after full course of vaccination
The endpoint of safety study | From the first dose of vaccination until 12 months after full course of vaccination
  Analysis of serious adverse events from the first dose of vaccination until 12 months after full course of vaccination

SECONDARY OUTCOMES:
The endpoint of efficacy study | Up to one year after the vaccination
  The number of severe and severity above COVID-19 cases 14 days after whole vaccination; The number of any severity of COVID-9 cases after first dose of vaccination; The number of COVID-19 cases of any severity in populations of different age group (18-59 years vs. 60 years and above) 14 days after whole vaccination.
Endpoint of immunogenicity and immune persistence study | At 14 days and 6 months after full course of vaccination
  The level of neutralizing antibody to SARS-COV-2 and IgG level of RBD protein binding antibody at 14 days and 6 months after full course of vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fangjun Li, Bachelor, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (18):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China
- Ecuador (3):
  - Biodimed Guayaquil Clinical Research Center, Guayaquil, Guayas
  - Biodimed Alemania Clinical Research Center, Quito, Pichincha
  - Biodimed Eloy Alfaro Clinical Research Center, Quito, Pichincha
- Indonesia (2):
  - Fkui-Rscm, Jakarta, Jakarta Special Capital Region
  - FK Unpad/RSHS, Bandung, West Java
- Pakistan (8):
  - Aziz Fatimah Hospital, Faisalabad, Punjab Province
  - Avicenna Hospital, Lahore, Punjab Province
  - Central Park Teaching Hospital, Lahore, Punjab Province
  - National Hospital & Medical Center, Lahore, Punjab Province
  - University of Health Sciences, Lahore, Punjab Province
  - Al-Shifa Trust Eye Hospital, Rawalpindi, Punjab Province
  - Indus Hospital and Health Network, Karachi, Sindh
  - Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad
- Uzbekistan (4):
  - Family Hospital No.15, Tashkent
  - GUVD Poliklinika, Tashkent
  - IIV Markaziy Poliklinika, Tashkent
  - Toshkent viloyat IIV Poliklinika, Tashkent

REFERENCES:
- [Derived] Dai L, Gao L, Tao L, Hadinegoro SR, Erkin M, Ying Z, He P, Girsang RT, Vergara H, Akram J, Satari HI, Khaliq T, Sughra U, Celi AP, Li F, Li Y, Jiang Z, Dalimova D, Tuychiev J, Turdikulova S, Ikram A, Flores Lastra N, Ding F, Suhardono M, Fadlyana E, Yan J, Hu Z, Li C, Abdurakhmonov IY, Gao GF; ZF2001 Global Trial Group. Efficacy and Safety of the RBD-Dimer-Based Covid-19 Vaccine ZF2001 in Adults. N Engl J Med. 2022 Jun 2;386(22):2097-2111. doi: 10.1056/NEJMoa2202261. Epub 2022 May 4. PMID 35507481